CLINICAL TRIAL: NCT03609476
Title: Trial of Void With Saline Bladder Instillation, a Randomized Controlled Trial
Brief Title: Trial of Void With Saline Bladder Instillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ronald Kaufman, MD (Other)
Responsible Party: Sponsor-Investigator, Ronald Kaufman, MD, Associate Professor of Surgery, Albany Medical College
Organization: Albany Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AMC4851
Record Dates: First submitted 2018-07-17; First posted 2018-08-01 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Urethral Catheter Removal After Urologic Procedure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care group (Active Comparator): No saline instillation
  Interventions: Procedure: No saline instillation
- Room temperature saline group (Active Comparator): room temperature saline instillation
  Interventions: Procedure: Room temperature saline instillation
- Warmed saline group (Active Comparator): warmed saline instillation
  Interventions: Procedure: Warmed saline instillation

INTERVENTIONS:
Procedure: Room temperature saline instillation — Saline is used as room temperature
  Arms: Room temperature saline group
Procedure: Warmed saline instillation — Saline is warmed to 37Celcius prior to instillation
  Arms: Warmed saline group
Procedure: No saline instillation — No saline is used prior to catheter removal
  Arms: Standard of care group

SUMMARY:
This study is being done to see if there is a difference between the traditional method of removing a urethral catheter after surgery and waiting for the patient to urinate on their own to the saline instillation method which places either room temperature or warmed saline into the patient's bladder through the catheter before removing the catheter.

DETAILED DESCRIPTION:
Voiding trials after surgery to remove a catheter can be done in different ways.

Traditional method: The catheter is removed and the patient will attempt to void.

Room temperature saline instillation: Room temperature saline will be placed in the patients bladder through the catheter. The catheter will be removed and the patient will attempt to void.

Warmed saline group: Saline that has been warmed to 37C will be placed in the patients bladder through the catheter. The catheter will be removed and the patient will attempt to void.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing trial of void after placement of indwelling urethral catheter after urologic procedure

Exclusion Criteria:

* Patient incontinent at baseline.
* Patient has chronic indwelling urinary catheter or uses clean intermittent catheterization at home.
* Patient has documented neurogenic bladder.
* No trained person to administer the instillation or perform consent.
* Patient refusal to participate.
* Patient unable to give informed consent.
* Patient is a prisoner.
* Patient is pregnant.
* Patient unable to participate in notifying nursing of voids.
* Nursing is unable to measure post void residual with bladder scan machine secondary to body habitus or other anatomical abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Time from catheter removal to determination of passing void trial | 6 hours
  The time from when the urinary catheter is removed to a successful voiding trial defined as Void of at least 100ml AND Post Void residual (PVR) <150 or <2/3 of the voided volume

SECONDARY OUTCOMES:
Catheter free rate | 30 days
  Subject questioned at 30 day follow up if required to have a catheter placed after leaving the hospital
Urinary tract infection free rate | 30 days
  Determined at 30 day phone call to patient
Post void residual (PVR) | Within 30 days
  Successful PVR is <150ml or <2/3 of the voided volume

CONTACTS AND LOCATIONS:
Overall Officials: Ronald P Kaufman, Jr., MD, Principal Investigator — Albany Medical College, Division of Urology
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Background] Emberton M, Fitzpatrick JM. The Reten-World survey of the management of acute urinary retention: preliminary results. BJU Int. 2008 Mar;101 Suppl 3:27-32. doi: 10.1111/j.1464-410X.2008.07491.x. PMID 18307683
- [Background] Boccola MA, Sharma A, Taylor C, Wong LM, Travis D, Chan S. The infusion method trial of void vs standard catheter removal in the outpatient setting: a prospective randomized trial. BJU Int. 2011 Apr;107 Suppl 3:43-6. doi: 10.1111/j.1464-410X.2011.10044.x. PMID 21492377
- [Background] Du J, Marshall D, Leyland J, Shaw L, Broome KE, Mason DF. Prospective, multicentre, randomized controlled trial of bladder filling prior to trial of void on the timing of discharge. ANZ J Surg. 2013 Apr;83(4):239-42. doi: 10.1111/j.1445-2197.2012.06253.x. Epub 2012 Sep 18. PMID 22984818
- [Background] Wilson ID, Bramwell SP, Hollins GW. A randomized trial comparing bladder infusion with standard catheter removal after transurethral resection of the prostate. BJU Int. 2000 Dec;86(9):993-5. doi: 10.1046/j.1464-410x.2000.00963.x. PMID 11119091
- [Background] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Lyth DR, Braslis K, Iacovou JW. The infusion trial of micturition. Br J Urol. 1997 Jan;79(1):94-5. doi: 10.1046/j.1464-410x.1997.30520.x. PMID 9043505
- [Background] Noble JG, Menzies D, Cox PJ, Edwards L. Midnight removal: an improved approach to removal of catheters. Br J Urol. 1990 Jun;65(6):615-7. doi: 10.1111/j.1464-410x.1990.tb14830.x. PMID 2372674
- [Background] Crowe H, Clift R, Duggan G, Bolton D, Costello A. Randomized study of the effect of midnight removal of urinary catheters. Urol Nurs. 1994 Mar;14(1):18-20. PMID 8153735
- [Background] Zimlichman E, Henderson D, Tamir O, Franz C, Song P, Yamin CK, Keohane C, Denham CR, Bates DW. Health care-associated infections: a meta-analysis of costs and financial impact on the US health care system. JAMA Intern Med. 2013 Dec 9-23;173(22):2039-46. doi: 10.1001/jamainternmed.2013.9763. PMID 23999949
- [Background] Richards MJ, Edwards JR, Culver DH, Gaynes RP. Nosocomial infections in combined medical-surgical intensive care units in the United States. Infect Control Hosp Epidemiol. 2000 Aug;21(8):510-5. doi: 10.1086/501795. PMID 10968716
- [Background] Klevens RM, Edwards JR, Richards CL Jr, Horan TC, Gaynes RP, Pollock DA, Cardo DM. Estimating health care-associated infections and deaths in U.S. hospitals, 2002. Public Health Rep. 2007 Mar-Apr;122(2):160-6. doi: 10.1177/003335490712200205. PMID 17357358
- [Background] Maki DG, Tambyah PA. Engineering out the risk for infection with urinary catheters. Emerg Infect Dis. 2001 Mar-Apr;7(2):342-7. doi: 10.3201/eid0702.010240. PMID 11294737
- [Background] Stenzelius K, Persson S, Olsson UB, Stjarneblad M. Noble metal alloy-coated latex versus silicone Foley catheter in short-term catheterization: a randomized controlled study. Scand J Urol Nephrol. 2011 Sep;45(4):258-64. doi: 10.3109/00365599.2011.560007. Epub 2011 Mar 31. PMID 21452931
- [Background] Gould CV, Umscheid CA, Agarwal RK, Kuntz G, Pegues DA; Healthcare Infection Control Practices Advisory Committee. Guideline for prevention of catheter-associated urinary tract infections 2009. Infect Control Hosp Epidemiol. 2010 Apr;31(4):319-26. doi: 10.1086/651091. No abstract available. PMID 20156062
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Tambyah PA, Oon J. Catheter-associated urinary tract infection. Curr Opin Infect Dis. 2012 Aug;25(4):365-70. doi: 10.1097/QCO.0b013e32835565cc. PMID 22691687
- [Background] Glynn A WV, Wilson J, et al. Hospital acquired infection: surveillance, policies and practice-a study of the control of hospital acquired infection in hospitals in England and Wales. In: Service PHL, ed. London1997.